CLINICAL TRIAL: NCT01963728
Title: Comparison of Insulin Isophane (NPH) With Insulin Glargine in New Onset Diabetes After Transplant (NODAT)
Brief Title: Comparison of Insulin Therapy in Treating Post-Transplant Diabetes
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Blood sugar status of the enrolled subjects wasn't evaluable
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Inova NODAT-001
Record Dates: First submitted 2013-10-10; First posted 2013-10-16 (Estimated); Results first posted 2022-01-12 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus
Keywords: post-transplant; diabetes mellitus; renal transplant; kidney transplant; lung transplant; heart transplant; insulin
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Insulin, Isophane; Isophane Insulin, Human; Insulin Glargine

STUDY DESIGN:
Masking Description: Subjects will be randomized to
  1. Insulin glargine (Lantus) or
  2. Insulin isophane (NPH)
Oversight: Data Monitoring Committee: No

ARMS (2):
- insulin isophane (Active Comparator): daily dose will be titrated based on fasting morning glucose values
  Interventions: Drug: Insulin, Isophane
- insulin glargine (Active Comparator): daily dose will be titrated based on fasting morning glucose values
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: Insulin, Isophane — daily dosing based on fasting morning glucose levels
  Other Names: human NPH
  Arms: insulin isophane
Drug: insulin glargine — daily dose based on fasting morning glucose levels
  Other Names: Lantus
  Arms: insulin glargine

SUMMARY:
To determine if the use of insulin isophane results in improved control of blood sugars compared to the use of insulin glargine in new onset diabetes after kidney, lung, or heart transplantation (NODAT).

DETAILED DESCRIPTION:
A large percentage of organ transplant recipients develop de novo diabetes mellitus after transplantation, also called "New Onset Diabetes After Transplant" or NODAT. The cause of the diabetes appears to be commonly used anti-rejection medications, particularly calcineurin inhibitors and glucocorticoids.

Management of glucose levels in NODAT often requires insulin therapy. Standard practice is to start long-acting insulin. However, patients with NODAT often exhibit fasting morning glucose levels that are relatively low compared to pre-lunch and pre-dinner glucose levels. This seems to make NODAT patients more susceptible to fasting, or morning, hypoglycemia on long-acting insulin analogues than non-transplant patients with type II diabetes. This phenomenon of morning hypoglycemia in NODAT often limits the up-titration of basal insulin resulting in suboptimal treatment of hyperglycemia later in the day. Because of this pattern, transplant patients may respond better to morning insulin isophane (intermediate acting) than to long-acting insulin glargine preparations.

Our trial is designed to compare morning NPH insulin (isophane insulin) with conventional therapy of basal glargine insulin on both continuous blood glucose levels and hemoglobin A1c (glycosylated hemoglobin).

ELIGIBILITY:
Inclusion Criteria:

1. Must be followed by the Inova Fairfax Hospital transplantation program for post-transplant care
2. Diabetes mellitus inadequately responsive to lifestyle modification and non-insulin hypoglycemic medication
3. Need for subcutaneous insulin therapy (after discontinuation of IV insulin therapy, if it was required)
4. Ability to read consent form and give consent in English.

Exclusion Criteria:

1. Use of insulin or non-insulin hypoglycemic medication before transplantation
2. Cystic fibrosis patients
3. Age < 18 years of age
4. Pregnancy
5. Non-English speaking subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-11-27 (Actual); Primary Completion 2015-04-09 (Actual); Study Completion 2015-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ross, MD, Principal Investigator — Inova Healthcare Services
Locations (1):
- Inova Fairfax Hospital, Falls Church, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
There is no data to share

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Medical Clinic
Period: Overall Study
Arm/Group | Insulin Isophane | Insulin Glargine
Started | 0 | 1
Completed | 0 (study terminated early) | 0 (study terminated early)
Not Completed | 0 | 1
Not completed — Study terminated early | 0 | 1

BASELINE CHARACTERISTICS:
Population: No patients enrolled in the insulin isophane arm
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Isophane | Insulin Glargine | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States |  | 1 | 1
basal insulin types administered [Number; unit: basal insulin type] — two types of basal insulin used in study
  basal insulin type |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin A1C (Glycosylated Hemoglobin)
Time Frame: at 6 months post enrollment
Population: study terminated early
Arm/Group | Insulin Isophane | Insulin Glargine
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Mean Blood Glucose Values
Description: measured by continuous glucose monitoring for 5 days
Time Frame: 3 and 6 months post enrollment
Population: No data study did not complete
Arm/Group | Insulin Isophane | Insulin Glargine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events collected over the 6 months each subject enrolled
Description: none reported
Arm/Group | Insulin Isophane | Insulin Glargine
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No